CLINICAL TRIAL: NCT03327935
Title: Malnutrition in Surgical Patients in the Faroe Islands: Post-discharge Nutrition and Resistance Training
Brief Title: Post-discharge Nutrition and Resistance Training in Surgical Patients
Acronym: MaSu
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Copenhagen (Other)
Collaborators: Health Insurance Fund of Research Council Faroe Islands (Unknown); National Hospital of the Faroe Islands (Other Government); Société des Produits Nestlé (SPN) (Industry)
Responsible Party: Principal Investigator, Jens Rikardt Andersen, Associate professor, University of Copenhagen
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: H-17000004
Record Dates: First submitted 2017-10-27; First posted 2017-11-01 (Actual); Last update posted 2020-07-23 (Actual); Status verified 2020-07

CONDITIONS: Malnutrition; Surgery
MeSH Terms: conditions — Malnutrition | interventions — Nutritional Status

STUDY DESIGN:
Intervention Model Description: 3 groups of 50 patients each by randomization
Masking Description: Baseline data are collected prior to the randomization and thus are masked. But during and after the intervention both participants and investigators are unblinded.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Nutrition (Experimental): Oral nutritional supplements and dietetic advice
  Interventions: Dietary Supplement: Nutrition
- Nutrition and exercise (Experimental): Oral nutritional supplements, dietetic advice and exercise training
  Interventions: Dietary Supplement: Nutrition
- Control (No Intervention): Standard Hospital Procedure

INTERVENTIONS:
Dietary Supplement: Nutrition — 150 Faroese surgical patients randomized to one of the following three arms 1) oral nutritional supplements and advice, 2) oral nutritional supplements and training exercise and 3) Standard hospital procedure. Primary outcome is loss of lean body mass
  Arms: Nutrition; Nutrition and exercise

SUMMARY:
Randomized intervention by nutritional supplements and training in postoperative patients after discharge

DETAILED DESCRIPTION:
Surgery combined with malnutrition is associated with loss of muscle mass and leads to serious consequences for the surgical patient. A majority of surgical patients continue to lose weight after discharge. Nutritional risk screening has not been fully implemented at Landssjúkrahúsið - the National Hospital of the Faroe Islands and therefore the prevalence of patients at nutritional risk is unknown. The aim of this study is to examine whether an intervention with independent nutritional supplements or an intervention combining nutritional supplements and resistance training is more effective in preventing loss of muscle mass than standard care in surgical patients following discharge. Secondary outcomes are changes in body weight, quality of life, muscle strength and activities of daily living. Furthermore, we want to screen hospitalized surgical patients for nutritional risk in order to get an estimate of the prevalence of nutritional risk.

ELIGIBILITY:
Inclusion Criteria:

* Admitted to the surgical departments at Landssjúkrahúsið - National Hospital of Faroe Islands
* Aged 18 years or above
* One or more of the following surgical procedures: knee alloplasty, hip alloplasty, collum femoris fracture, back fracture, abdominal surgery, mamma surgery and other comprehensive surgery
* At nutritional risk according to screening

Exclusion Criteria:

* Minimally invasive surgery/Laparoscopic surgery
* Severely reduced kidney function (p-creatinin>250 mikromol/l) or dialysis
* Terminal illness
* Inability to cooperate in tests or exercises due to cognitive function or dementia
* Admitted to intensive care unit
* Inability to speak or understand Faroese, Danish or English
* Consent according to national regulations not obtainable

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2018-05-01 (Actual); Primary Completion 2020-04-01 (Actual); Study Completion 2020-04-01 (Actual)

PRIMARY OUTCOMES:
Loss of lean body mass | 8 weeks
  Non-bone lean mass measured by dual energy x-ray absorptiometry (DXA) whole-body scans

CONTACTS AND LOCATIONS:
Overall Officials: Jens Rikardt R Andersen, Study Chair — University of Copenhagen
Locations (1):
- National Hospital of Faroe Islands, Tórshavn, Faroe Islands

IPD SHARING:
Plan to Share IPD: No